CLINICAL TRIAL: NCT02075658
Title: A Comparative Study of the Physiological Response, Between AirSeal, an Integrated Insufflation and Access System, and Conventional Insufflation and Trocars
Brief Title: A Comparative Study Between AirSeal, an Integrated Insufflation System, and Conventional Insufflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jaime Landman, Professor of Urology and Radiology Chairman, Department of Urology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012-9088
Record Dates: First submitted 2013-11-01; First posted 2014-03-03 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; minimally invasive procedures; robotic nephrectomy; laparoscopic nephrectomy; pneumoperitoneum; trocars; AirSeal® IFS
MeSH Terms: conditions — Carcinoma, Renal Cell; Pneumoperitoneum | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Insufflation and Trocars (Other): Subjects enrolled in this study arm will have their procedure performed using either the conventional insufflator and trocars. This system have been cleared for use by the FDA's 510 (k)process and are currently employed in clinical practice, including at UC Irvine Medical Center.
  Interventions: Device: Conventional Insufflator and Trocar
- AirSeal® System-Interventional (Active Comparator): The AirSeal® System consists of an insufflation, filtration, and recirculation system (AirSeal® IFS), a triple lumen filtered tube set, and a valve free trocar (AirSeal® Access Port).
  Interventions: Device: AirSeal® System-Interventional

INTERVENTIONS:
Device: AirSeal® System-Interventional — The AirSeal® System consists of an insufflation, filtration, and recirculation system (AirSeal® IFS), a triple lumen filtered tube set, and a valve free trocar (AirSeal® Access Port). The device enables peritoneal access with a novel mechanism to maintain pneumoperitoneum without a mechanical seal.
  Arms: AirSeal® System-Interventional
Device: Conventional Insufflator and Trocar — Conventional insufflator and trocars are used in standard procedures and will serve as the base for comparison of the study device (AirSeal® System).
  Arms: Conventional Insufflation and Trocars

SUMMARY:
Renal cancer has traditionally been treated by surgical removal of the tumor, as the tumors are resistant to chemotherapy and radiation. The traditional treatment, where the entire kidney and tumor were removed through an abdominal incision, may now have more long term problems than the actual cancer. As a result, less invasive techniques have been developed such as laparoscopic surgery where the abdomen is inflated with carbon dioxide (i.e. via an insufflation system) and the surgery performed with special instruments through small ports, known as trocars. Rapid advances in minimally invasive surgical techniques demand ongoing technological improvement.

Conventional insufflators and trocars allow for laparoscopic surgery to occur, however the system does not account for pressure changes within the abdomen when instruments are inserted or removed. The AirSeal® System consisting of an insufflation, filtration, and recirculation system (AirSeal® IFS), a triple lumen filtered tube set, and a valve free trocar (AirSeal® Access Port) has been designed to create and maintain the pressure barrier throughout the procedure. The objective of this study is to collect comparative physiological, pulmonary compliance and surgical utility data for both the AirSeal® System and conventional insufflators and trocars in a controlled population undergoing laparoscopic/robotic renal or peri-renal procedures. Subjects enrolled in this study will have their procedure performed using either the AirSeal® System or a conventional insufflator and trocars. Both systems have been cleared for use by the FDA's 510(k) process and are currently employed in clinical practice, including at University of California, Irvine Medical Center. We hypothesize that with the use of the AirSeal® System, laparoscopic efficiencies and outcomes will be significantly greater than with the conventional insufflator and trocars system.

DETAILED DESCRIPTION:
Rapid advances in minimally invasive surgical techniques demand ongoing technological improvement.

The benefits of laparoscopic surgery to patient comfort and recovery have been made with procedures such as the cholecystectomy and gastric bypass. The AirSeal® System consists of an insufflation, filtration, and recirculation system (AirSeal® IFS), a triple lumen filtered tube set, and a valve free trocar (AirSeal® Access Port). The device enables peritoneal access with a novel mechanism to maintain pneumoperitoneum without a mechanical seal. Specifically, the AirSeal® System creates a pressure barrier within the proximal housing of the cannula which acts as an invisible seal to maintain pneumoperitoneum during the course of surgery. It utilizes a re-circulation and filtration control unit (AirSeal® IFS) designed specifically for the AirSeal® Access Port to create and maintain the pressure barrier. The AirSeal® System has applications in abdominal minimally invasive surgical procedures to establish a path of entry for laparoscopic instruments. The insufflation and recirculation system (AirSeal® IFS) is reusable and the AirSeal® Access Port and triple lumen filtered tube set are designed as single patient use devices. The 1st generation AirSeal® System received FDA 510(k) clearance in 2007 and the current system received FDA 510(k) Clearance in May 2011. Since that time, the AirSeal™ system has been used routinely in centers throughout the United States and has been observed by surgeons and anesthesia teams to provide a more gentle, stable, and consistent pneumoperitoneum. Initial evidence of this has reported in the literature1. Kavoussi and colleagues state; "We have found that patients had blunted end-tidal carbon dioxide (CO2) levels and CO2 elimination rates compared with the CO2 elimination rates observed in studies evaluating transperitoneal laparoscopy using the conventional trocar. To determine if a difference truly exists, CO2 elimination rates must be prospectively analyzed in a head to head comparison between valve-less and conventional trocars." This study is designed to compare the physiological impact and pulmonary compliance of patients undergoing laparoscopic/robotic renal or peri-renal surgery with and without the AirSeal® System.

1 A new Valve-Less Trocar for Urology Laparoscopy: Initial Evaluation. Journal of Endourology 2009;23: 1535-39

ELIGIBILITY:
Inclusion Criteria:

1. Competent adult (18 years of age and older) males and females.
2. Persons undergoing laparoscopic/robotic renal or peri-renal procedures.

Exclusion criteria:

1. Under age 18
2. Unable to provide informed consent
3. Have a history of ascites
4. History of transplant kidney
5. Solitary kidney (one kidney)
6. Uncontrolled Diabetes (HbA1c > 8)
7. Pregnancy (as noted by standard of care history and physical)
8. Women who are breast-feeding
9. History of narcotic abuse or chronic pain
10. Emergency Surgery
11. Person's participating in any other research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-01; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bucur P, Hofmann M, Menhadji A, Abedi G, Okhunov Z, Rinehart J, Landman J. Comparison of Pneumoperitoneum Stability Between a Valveless Trocar System and Conventional Insufflation: A Prospective Randomized Trial. Urology. 2016 Aug;94:274-80. doi: 10.1016/j.urology.2016.04.022. Epub 2016 Apr 27. PMID 27130263

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Competent adults (>18 years old)(male or female) undergoing laparoscopic/robotic renal or peri-renal procedures will be included in this study.
Period: Overall Study
Arm/Group | Conventional Insufflation and Trocars | AirSeal® System-Interventional
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Insufflation and Trocars | AirSeal® System-Interventional | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (13.1) | 62.5 (15.3) | 63.7 (28.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 18 | 23 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 24 | 22 | 46
  Black | 1 | 1 | 2
  Asian | 1 | 2 | 3
  Hawaiian/PI | 0 | 1 | 1
  Other | 2 | 2 | 4
Charlson Comorbidity Index [Mean (Standard Deviation); unit: units on a scale (0-43)] — 0 = no comorbidities, minimal chance of mortality 43 = many comorbidities, very high chance of mortality CCI predicts a patients 10 year mortality rate based on comorbidities
  units on a scale (0-43) | 3.2 (1.7) | 3.6 (2.4) | 3.4 (2.1)
Treatment [Count of Participants; unit: Participants]
  Radical Nephrectomy | 8 | 9 | 17
  Simple Nephrectomy | 1 | 0 | 1
  Partial Nephrectomy | 11 | 9 | 20
  Nephroureterectomy | 1 | 3 | 4
  Cryoablation | 5 | 4 | 9
  Pyeloplasty | 1 | 2 | 3
  Ureteral implantation | 0 | 1 | 1
  Retroperitoneal mass excision | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: AirSeal Reduction in the Variance of Intra-abdominal Pressure
Description: Our primary aim is to show reduction in the variance of intra-abdominal pressure throughout the operative procedure when using the AirSeal device compared to a conventional insufflator. Based on preliminary data, we assume pressures maintained at a mean of 15 through out surgery for both devices and a variance of 3.6 with the conventional insufflator.
Time Frame: Day 1 (Day of Procedure)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conventional Insufflation and Trocars | AirSeal® System-Interventional
Number analyzed (Participants) | 28 | 28
mmHg | 5.5 (3.3) | 1.3 (1.1)

2. Secondary Outcome: Improvement in Cardiac Output With the AirSeal Device.
Description: Assuming cardiac output of approximately 5.0 L/min with the conventional device, we will have 96% power to detect as significant an improvement in cardiac output to 5.5 L/min using a two-group Satterwaite t-test and assuming variance of 0.25.
  Cardiac out put is defined by the volume of blood pumped by the heart in a given amount of time.
Time Frame: Day 1 (Day of Procedure)
Measure: Mean (Standard Deviation); unit: volume per minute
Arm/Group | Conventional Insufflation and Trocars | AirSeal® System-Interventional
Number analyzed (Participants) | 28 | 28
volume per minute | NA (NA) — Current staff is unable to locate the analysed data from the original study and only has the published article to go by. We do not have the mean and standard deviation for this outcome measure. We only have the interpreted results from the paper. | NA (NA) — Current staff is unable to locate the analysed data from the original study and only has the published article to go by. We do not have the mean and standard deviation for this outcome measure. We only have the interpreted results from the paper.

ADVERSE EVENTS:
Arm/Group | Conventional Insufflation and Trocars | AirSeal® System-Interventional
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No